CLINICAL TRIAL: NCT03055221
Title: TRUST-2: An Open-label Continuation Trial of the Safety and Efficacy of Intravenous Remodulin® in Patients in India With Pulmonary Arterial Hypertension (PAH)
Brief Title: TRUST-2: Safety and Efficacy of Intravenous Remodulin® in Patients in India With Pulmonary Arterial Hypertension (PAH)
Acronym: TRUST-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIV-PH-403
Record Dates: First submitted 2017-02-09; First posted 2017-02-16 (Actual); Results first posted 2017-07-28 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Remodulin; 6-Minute Walk Test
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intravenous Treprostinil (Experimental): Intravenous treprostinil was supplied as 1 mg/mL.
  Interventions: Drug: Intravenous Treprostinil

INTERVENTIONS:
Drug: Intravenous Treprostinil — Intravenous treprostinil supplied in 20-mL vials and diluted to the appropriate concentration for administration.
  Other Names: Remodulin

SUMMARY:
This was an open-label extension of Study RIV-PH-402, TRUST-1: Treprostinil for Untreated Symptomatic Pulmonary Arterial Hypertension (PAH) Trial. Subjects who completed Study RIV-PH-402 were eligible to enroll.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were enrolled in and completed Study RIV-PH-402 (TRUST-1)

Exclusion Criteria:

* Subjects who were unblinded for potential rescue therapy in Study RIV-PH-402 and were found to be allocated to the Remodulin treatment group were not eligible to participate in this study.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-06-10 (Actual); Primary Completion 2014-02-25 (Actual); Study Completion 2014-02-25 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous Treprostinil: Intravenous treprostinil was supplied as 1 mg/mL.
  Remodulin (Intravenous Treprostinil): Intravenous treprostinil supplied in 20-mL vials and diluted to the appropriate concentration for administration.
Period: Overall Study
Arm/Group | Intravenous Treprostinil
Started | 20
Completed | 0
Not Completed | 20
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 4
Not completed — Death | 6
Not completed — Physician Decision | 1
Not completed — Study terminated by Sponsor | 3
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Intravenous Treprostinil
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  India | 16

OUTCOME MEASURES:

1. Primary Outcome: Effect of Long-term Remodulin Therapy on the 6-Minute Walk Distance (6MWD)
Description: The intent of the 6-Minute Walk Test (6MWT) is to evaluate exercise capacity associated with carrying out activities of daily living.
Time Frame: The 6MWD was assessed at each subject's last visit, which occurred up to approximately 9 years after first visit
Population: Data are presented for subjects who completed the 6MWT at their final visit. Not all subjects completed a 6MWT at their final visit.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Intravenous Treprostinil
Number analyzed (Participants) | 13
Meters | 440.8 (108.6)

2. Primary Outcome: Effect of Long-term Remodulin Therapy on the NYHA Functional Classification
Description: The NYHA functional classification ranges from I (subject's disease does not affect daily activities) to IV (subject's disease causes severe impairment).
Time Frame: The NYHA functional classification was assessed at each subject's last visit, which occurred up to approximately 9 years after first visit
Population: Data presented include all subjects who underwent an NYHA functional classification assessment at their final visit. Not all subjects underwent an NYHA assessement at their final visit.
Measure: Mean (Standard Deviation); unit: Functional Class
Arm/Group | Intravenous Treprostinil
Number analyzed (Participants) | 11
Functional Class | 2.1 (0.6)

3. Primary Outcome: Effect of Long-term Remodulin Therapy on Subject Safety
Description: Safety was assessed by summarizing the number of subjects with at least 1 AE during the 12 weeks (or until premature termination).
Time Frame: Baseline to Week 12
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Treprostinil
Number analyzed (Participants) | 16
Participants | 14

ADVERSE EVENTS:
Time Frame: Baseline to each subject's last visit, assessed up to approximately 9 years.
Arm/Group | Intravenous Treprostinil
All-Cause Mortality (participants affected / at risk) | 6/16
Serious Adverse Events (participants affected / at risk) | 14/16
Other Adverse Events (participants affected / at risk) | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Treprostinil (N=16)
Bacteraemia (Infections and infestations) | 2 (2)
Pyrexia (General disorders) | 5 (5)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Catheter site swelling (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Device dislocation (General disorders) | 3 (5)
Disease progression (General disorders) | 1 (1)
Infusion site pain (General disorders) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 4 (5)
Device-related infection (Infections and infestations) | 3 (3)
Device-related sepsis (Infections and infestations) | 2 (2)
Endocarditis (Infections and infestations) | 1 (1)
Localized infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (2)
Nasopharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Polymenorrhea (Reproductive system and breast disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abortion induced (Surgical and medical procedures) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Treprostinil (N=16)
Cyanosis (Cardiac disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (5)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Local swelling (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (3)
Catheter site pain (General disorders) | 3 (5)
Wound infection (Infections and infestations) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Weight decreased (Investigations) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (5)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Gynacomastia (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Right ventricular failure (Cardiac disorders) | 1 (1)
Chills (General disorders) | 1 (3)
Device dislocation (General disorders) | 1 (1)
Catheter site swelling (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any interim results of the Study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.